CLINICAL TRIAL: NCT00752778
Title: MRI Follow-up of Macrophagic Infiltration in MS Patients Treated With Tysabri
Brief Title: Magnetic Resonance Imaging (MRI) Follow-up of Macrophagic Infiltration in MS Patients Treated With Tysabri
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4118
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Multiple Sclerosis
Keywords: MRI, PET scan
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: pet-scan FDG-F18

SUMMARY:
To evaluate the diagnosis value of MRI and positon emission tomography (PET) scan for studying macrophagic infiltration and other brain modification in multiple sclerosis (MS) patients treated with Natalizumab (Tysabri).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with MS
* Treatment with Tysabri planned

Exclusion Criteria:

* Allergy to Tysabri or MRI contrast products
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Number of enhanced lesions on MRI before and after treatment. PET scan modification in brain (in enhanced lesions and in the whole brain). | At baseline and after 3 months of treatment.

SECONDARY OUTCOMES:
Correlation with relapses. | During the 3 months of treatment and the 3 following months.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme DE SEZE, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (3):
- France (3):
  - Service de Neurologie, Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service de Médecine Nucléaire, Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service de Radiologie 2, Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg